CLINICAL TRIAL: NCT03149913
Title: Does Local Paclitaxel Improve the Efficacy of Balloon Angioplasty Without Stent Implantation for Treatment of Below the Knee Artery Lesions?
Brief Title: Local Paclitaxel or Balloon Angioplasty Below the Knee
Acronym: SAMBA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Dr. med. Gunnar Tepe (Other)
Collaborators: InnoRa GmbH (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Gunnar Tepe, Director of the Deparment of Radiology, Clinical Professor, Klinikum Rosenheim
Organization: Klinikum Rosenheim (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTK 1
Record Dates: First submitted 2017-03-30; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Stenosis; Occlusion; Restenosis
Keywords: below the knee artery; endovascular; drug coated balloon; critical limb ischemia
MeSH Terms: conditions — Constriction, Pathologic; Bites and Stings; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: The vessel patency (measured by angiography at 6 months) will be compared after patients have been treated either with paclitaxel coated or uncoated balloons (control) in BTK arteries
Who Masked: Participant
Masking Description: drug coated balloon versus uncoated balloon
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug coated balloon (Experimental): SeQuentPlease OTW paclitaxel coated balloon catheter
  Interventions: Device: SequentPlease OTW paclitaxel coated balloon catheter
- uncoated PTA balloon catheter (Active Comparator): Standard of care uncoated BTK balloon catheter
  Interventions: Device: conventional uncoated balloon for BTK endovascular therapy

INTERVENTIONS:
Device: SequentPlease OTW paclitaxel coated balloon catheter — PTA with SequentPlease OTW paclitaxel coated balloon catheter
  Arms: Drug coated balloon
Device: conventional uncoated balloon for BTK endovascular therapy — PTA with uncoated balloon for BTK endovascular therapy
  Arms: uncoated PTA balloon catheter

SUMMARY:
Patients with claudication or critical limb ischemia will be treated either with uncoated balloons or paclitaxel coated balloons in order to enhance the vessel patency in stenosed or occluded below the knee arteries

DETAILED DESCRIPTION:
After successful guide wire passage of the below the knee index lesions the patients will either receive a treatment with a conventional uncoated balloon or a balloon coated with paclitaxel. Only patients who require follow-up angiography after 6 months will be included in this study. The primary endpoint (index vessel occluded or still open) is at 6 months - the patients will be also followed for 24 months for clinical endpoints. In addition an MRI is planned at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Chronic stenotic or occlusive atherosclerotic disease of the infrapopliteal arteries
* Rutherford 2-5 patients
* Patients with ≤ 2 BTK lesions (≥ 70% diameter stenosis)
* Lesion length limited to 5-25 cm

Exclusion Criteria:

* Planned or foreseeable amputation
* Previous amputation at the index limb
* Index vessel with no run-off to the foot distal to the index lesion
* Prior treatment of the index lesion with a drug coated balloon
* In-stent restenosis
* Life expectancy <1 year
* Known creatinine >1.4 mg% if patient is not on dialysis
* Acute thrombus in the index limb
* Aneurysm in the index leg
* Known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, abciximab, paclitaxel
* Patients with concomitant medical illnesses that require cytostatic or radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Occlusion rate of the target lesion at 6 months | 6 +/- 1 months
  by digital substraction angiogram or MRI

SECONDARY OUTCOMES:
target lesion revascularization | 3, 6, 12 and 24 months
  repeat intervention

OTHER OUTCOMES:
Walking distance | 3, 6, 12 and 24 months
  Evaluation of Rutherford category
Wound status | 3, 6, 12 and 24 months
  improvement, no change, worsening

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tepe, MD, Principal Investigator — RoMed Klinikum Rosenheim
Locations (7):
- LKH-Univ. Klinikum Graz, Graz, Austria
- Germany (6):
  - Herzzentrum Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - Tepe, Rosenheim, Baden-Wurttemberg
  - Klinikum Arnsberg, Arnsberg
  - Ev.-Luth. Diakonissenanstalt zu Flensburg, Flensburg
  - Evangelisches Krankenhaus Mülheim a. d. Ruhr, Mülheim
  - Universitätsklinikum Würzburg, Würzburg